CLINICAL TRIAL: NCT01435564
Title: Innovations in Mobile Phone Based Physical Activity- A Pilot of Clinical Trial in Sedentary Men and Women
Brief Title: Pilot Study: Mobile Phone Based Physical Activity in Sedentary Men and Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Heart Association (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P0030018; K23NR011454 (NIH)
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Sedentary Lifestyle; Physical Activity
Keywords: Mobile phone; Sedentary lifestyle; Physical activity; Prevention; Health Promotion; Exercise; eHealth; Electronic diary
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pedometer (Active Comparator)
  Interventions: Behavioral: pedometer only
- Mobile phone physical activity intervention (Experimental)
  Interventions: Behavioral: Mobile phone

INTERVENTIONS:
Behavioral: Mobile phone — Participants in this group will receive both the pedometer and the mobile-phone based physical activity intervention fot three months.
  Other Names: Mobile phone based physical activity intervention
  Arms: Mobile phone physical activity intervention
Behavioral: pedometer only — Participants in this group will receive only a pedometer.
  Arms: pedometer

SUMMARY:
The purpose of this pilot study is to estimate the efficacy of a mobile phone based physical activity intervention in sedentary men and women.

ELIGIBILITY:
Inclusion Criteria:

1. Sedentary lifestyle at work and/or during leisure time
2. Male or female, age between 21-69
3. Access to a telephone at home or a mobile phone
4. Speak and read English
5. BMI between 20-43 kg/m2

Exclusion Criteria:

1. Known medical condition or other physical problems that need special attention in an exercise program
2. Planning a trip out of the United States during the study
3. Pregnant/Delivered a baby during the last 6 months
4. HIV positive
5. Known severe hearing or speech problems
6. Currently participating in lifestyle modification programs or research studies (such as physical activity, diet, and/or weight loss programs)

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Pedometer measured steps | 3 months

SECONDARY OUTCOMES:
7-Day Physical Activity Recall | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yoshimi Fukuoka, PhD, RN, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States